CLINICAL TRIAL: NCT04623164
Title: Efficacy of Complex Phytoadaptogenes as an Adjunct to Non-surgical Periodontal Treatment in Patients With Chronic Periodontitis: a Randomized Clinical Trial
Brief Title: Complex Phytoadaptogenes in Chronic Periodontitis Treatment.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vladikavkaz Scientific Center of the Russian Academy of Sciences (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Interventional 24.01.2019
Record Dates: First submitted 2020-10-20; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-10

CONDITIONS: Chronic Periodontitis
Keywords: complex phytoadaptogenes; periodontitis; periodontal pathogens; microcirculation; Glycyrrhiza glabra; Rhodiola rosea; Acantopanax senticosus
MeSH Terms: conditions — Chronic Periodontitis; Periodontitis | interventions — Glycyrrhiza glabra extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 Group (Control) (No Intervention): ten students with healthy periodontium
- 2 Group (Experimental): ten patients receiving standard non-surgical periodontal treatment (NSPT)
  Interventions: Procedure: Standard non-surgical periodontal treatment (NSPT)
- 3 Group (Experimental): ten patients receiving standard non-surgical periodontal treatment NSPT + 28-day chronotherapy with complex phytoadaptogens (CFA)
  Interventions: Drug: Cocktail from complex phytoadaptogens (CFA); Procedure: Standard non-surgical periodontal treatment (NSPT)

INTERVENTIONS:
Drug: Cocktail from complex phytoadaptogens (CFA) — Cocktail from complex phytoadaptogens (CFA) is composed from 70% alcohol extracts of Glycyrrhiza glabra, Rhodiola rosea, Acantopanax senticosus in the ratio 2:1:1. Application of CFA in 3 group was carried out after non-surgical periodontal therapy (NSPT). After NSPT the patient filled out an Estberg questionnaire to determine the chronotype. After processing the questionnaire, a chronotype was identified and the patient was prescribed CFA dosage. Application of CFA was carried out in the periods of exacerbation of chronic periodontitis within 28 days with a dosage of CFA depending on the chronotype of the person - morning chronotype at 45 drops in the morning before 10.00 o'clock; independent chronotype 20 drops 3 times a day; evening chronotype 30 drops at 14.00 o'clock and 20 drops at 19.00 o'clock.
  Other Names: Glycyrrhiza glabra, Rhodiola rosea, Acantopanax senticosus
  Arms: 3 Group
Procedure: Standard non-surgical periodontal treatment (NSPT) — Oral hygiene instructions (including brushing technique, the use of interdentally flosses, and/or brushes), NSPT (mouth scaling and root planing using an ultrasonic scaler UDS-L LED (Woodpecker, China) and Graceys curettes (Hu Friedy, Chicago, USA)). The treated periodontal pockets were irrigated with 0.12% chlorhexidine gluconate. Patients were given recommendation to rinse their mouth three times daily for 14 days using 0.12% chlorhexidine gluconate
  Arms: 2 Group; 3 Group

SUMMARY:
A randomized controlled clinical trial was done to assess the periodontal status of the individuals baseline followed by by including chronotherapy with complex phytoadaptogens (CFA) into the non-surgical periodontal treatment (NSPT). The periodontal parameters were again assessed after and compared with the control group (participants with healthy periodontium) and group with non-surgical periodontal treatment (NSPT).

DETAILED DESCRIPTION:
The aim of this study was to increase the effectiveness of treatment and prevention of chronic generalized periodontitis and increase remission periods by including chronotherapy with complex phytoadaptogens (CFA) into the non-surgical periodontal treatment (NSPT).

Methods: Thirty systemically healthy patients, who had generalized chronic periodontitis with probing pocket depth (PPD) ≥5 mm, plaque index score <1,5 and the ability to maintain optimum oral hygiene after the initial phase of treatment, were included in the present investigation. Patients were divided into 3 groups: 1 Group - control (10 students with healthy periodontium); 2 Group - 10 patients receiving standard non-surgical periodontal treatment (NSPT); 3 Group - CFA application (10 patients receiving NSPT + 28-day chronotherapy with complex phytoadaptogens (CFA)). Control examinations were carried out in the following periods: before, after and 6 months after treatment. After each study time point the patients were able to visit the dental office to assess the periodontal status. The examination included the following:

1. Estberg questionnaire to determine the chronotype once before treatment;
2. Simplified Oral Hygiene Index John C. Greene Jack R. Vermillion (1964) (OHI-S);
3. Sulcus Bleeding Index Muhleman. H.R (1975) (SBI);
4. Periodontal Index Rusell. A.L (1956) (PI);
5. Doppler ultrasound. Patients of 2 and 3 groups received oral hygiene instructions (including brushing technique, the use of interdentally flosses, and/or brushes), NSPT (mouth scaling and root planing using an ultrasonic scaler UDS-L LED (Woodpecker, China) and Graceys curettes (Hu Friedy, Chicago, USA)). The treated periodontal pockets were irrigated with 0.12% chlorhexidine gluconate. Patients were given recommendation to rinse their mouth three times daily for 14 days using 0.12% chlorhexidine gluconate Statistical Analysis: Statistical analyses were performed using Statistica 10,0 software ("StatSoft, Inc", Russia). Data were investigated by nonparametric method with determination of median (Md) and interquantile ranges (25th and 75th percentile) due to the small number of variants in the sample (Wilcoxon test). Data were compared before, after and 6 months after treatment. Statistically significant differences in all statistical tests was set to P<0.05.

ELIGIBILITY:
Inclusion Criteria:

* the presence of chronic periodontitis with probing pocket depth (PPD) ≥5 mm, plaque index score <1,5; age from 20-45 years; according to the patients, there is no somatic pathology

Exclusion Criteria:

* age younger than 20 and older than 45 years; diabetes; chronic somatic diseases; infectious diseases; malignant neoplasms of various organs and systems; viral infections; autoimmune diseases; mental illness; pregnancy and lactation in women

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Periodontal Index Rusell. A.L (1956) | 6 months
  Changes in clinical parameter PI (Periodontal Index Rusell. A.L (1956)) in chronic periodontitis patients of group 2 (with NSPT) and group 3 (NSPT + 28-day use of CFA) from baseline to 6 months.
  Index shows severity of gingivitis, the presence of periodontal pockets, tooth mobility and alveolar bone loss. Evaluation of results: 0.1 - 1.5 points - I stage; 1.5 - 4.0 points - stage II; 4.0 - 8.0 points - stage III.
Sulcus Bleeding Index Muhleman. H.R (1975) (SBI) | 6 months
  Changes in clinical parameter SBI (Sulcus Bleeding Index Muhleman. H.R (1975)) in chronic periodontitis patients of group 2 (with NSPT) and group 3 (NSPT + 28-day use of CFA) from baseline to 6 months.
  Index is used for assessment of gingival bleeding. Evaluation of results: score 0 - gingival of normal texture and color, no bleeding; score 1 - gingival apparently normal, bleeding on probing; score 2 - bleeding on probing, change in color, no oedema; score 3 - bleeding on probing change in color, slight oedema; score 4 - either: (a) bleeding on probing, change in color, obvious oedema; or (b) bleeding on probing, obvious oedema; score 5 - bleeding on probing and spontaneous bleeding, change in color, marked oedema.

SECONDARY OUTCOMES:
Systolic flow velocity (S) | 6 months
  Systolic flow velocity (S) (Vad, mm/sec) was investigated by Doppler ultrasound in chronic periodontitis patients of group 2 (with non-surgical periodontal therapy (NSPT)) and group 3 (NSPT + 28-day use of complex phytoadaptogens (CFA)) from baseline to 6 months
Diastolic flow velocity (D) | 6 months
  Diastolic flow velocity (D) (Vad, mm/sec) was investigated by Doppler ultrasound in chronic periodontitis patients of group 2 (with non-surgical periodontal therapy (NSPT)) and group 3 (NSPT + 28-day use of complex phytoadaptogens (CFA)) from baseline to 6 months
Medium flow velocity (M) | 6 months
  Medium flow velocity (M) (Vad, mm/sec) was investigated by Doppler ultrasound in chronic periodontitis patients of group 2 (with non-surgical periodontal therapy (NSPT)) and group 3 (NSPT + 28-day use of complex phytoadaptogens (CFA)) from baseline to 6 months
Pulsatory index Gosling (PI) | 6 months
  Pulsatory index Gosling (PI) (relevant units) - reflects the elastic properties of the arteries; was investigated by Doppler ultrasound in chronic periodontitis patients of group 2 (with non-surgical periodontal therapy (NSPT)) and group 3 (NSPT + 28-day use of complex phytoadaptogens (CFA)) from baseline to 6 months
Resistance index (RI) | 6 months
  Resistance index (RI) (relevant units) - reflects the state of blood flow resistance distal to the measurement site; was investigated by Doppler ultrasound in chronic periodontitis patients of group 2 (with non-surgical periodontal therapy (NSPT)) and group 3 (NSPT + 28-day use of complex phytoadaptogens (CFA)) from baseline to 6 months
Stuart index (SD) | 6 months
  Stuart index (SD) (relevant units) - reflects the elastic properties of the arteries; was investigated by Doppler ultrasound in chronic periodontitis patients of group 2 (with non-surgical periodontal therapy (NSPT)) and group 3 (NSPT + 28-day use of complex phytoadaptogens (CFA)) from baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Datieva, M.D., Principal Investigator — Vladikavkaz Scientific Centre of Russian Academy of Sciences
Locations (1):
- 1Institute of Biomedical Investigations - the Affiliate of Vladikavkaz Scientific Centre of Russian Academy of Sciences, Vladikavkaz, RSO-Alania, Russia

IPD SHARING:
Plan to Share IPD: No